CLINICAL TRIAL: NCT04036695
Title: Investigation of Electrophysiological Substrate of Arrhythmia in Hemodialysis Patients
Brief Title: Arrhythmia in Hemodialysis Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Chris McIntyre, Professor of Medicine, Medical Biophysics, and Paediatrics, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 113905
Record Dates: First submitted 2019-07-17; First posted 2019-07-30 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Arrythmia, Cardiac; Sudden Cardiac Death; Hemodialysis
MeSH Terms: conditions — Arrhythmias, Cardiac; Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Reveal LINQ insertable cardiac monitoring system (Experimental): In this all study, participants will have the option to undergo an insertion procedure of the Reveal LINQ insertable cardiac monitoring system on a dialysis or non-dialysis treatment day at University Hospital. The implantable loop recorder will be monitored at least once a week for up to 12 months.
  Interventions: Device: Reveal LINQ insertable cardiac monitoring system

INTERVENTIONS:
Device: Reveal LINQ insertable cardiac monitoring system — A small implantable cardiac monitor (Reveal LINQ device) will be inserted under local anaesthetic in an outpatient procedure. The Reveal LINQ device is composed of two electrodes and is used to continuously monitor electric activity temporally. It can detect arrhythmic episode and record up to 27 minutes of electrocardiographic (ECG) activity. This device is capable of continuous monitoring of patient's ECG activity for up to three years and will be utilized in this study to obtain initial information on the timing and nature of the arrhythmia suffered by hemodialysis patients leading to SCD.

SUMMARY:
Patients receiving dialysis for kidney failure suffer from very high rates of sudden cardiac death due to abnormal heart rhythms and perfusion defects associated with HD treatment. It has previously been recognized that patients suffer heart injury during the dialysis procedure which may be an important factor for investigation. The study uses a simple implantable device that can monitor heart rhythms over time to gather information on the type of abnormal rhythms that occur in dialysis patients. This information will be combined with ultrasound and x-ray scans of the heart that will also be collected. The goal is to understand the relationship between the abnormal rhythms and injury to the heart during dialysis and what causes these injuries. The information gathered in this study will be used to compare the accuracy of an in house personalized computational model to predict potential cardiac injuries when patients undergo HD treatment.

DETAILED DESCRIPTION:
This is an exploratory, single group, observational study involving patients recruited from the dialysis patient population of the London Health Science Centre (LHSC) Regional Renal Program. Recruited patients will undergo insertion of the Reveal LINQ insertable cardiac monitoring system and will continuously be examined over a time period of up to 12 to 24 months to gather data on the incidence of arrhythmia.

Those patients enrolled into the study will have their first study session on their midweek dialysis treatment day (Wednesday or Thursday) at St. Joseph's Hospital. During the first study visit, all participants will have an external multichannel ECG, CT scan, CT angiogram, and 2D echo done. In addition to this, all participants will have non-invasive monitoring of circulatory stress using the CVInsight contact device, and blood work will be drawn. Within one month, all participants will have a second study visit where they will undergo the same study procedures as in session one with the addition of up to 30 minutes of intradialytic exercise. This visit will also take place at St. Joseph's Hospital on a mid-week dialysis treatment day. If a patient would like to, they will then undergo an insertion procedure of the Reveal LINQ insertable cardiac monitoring system on a dialysis or non-dialysis treatment day at University Hospital. Dr. Allan Skanes (CoInvestigator) will perform this procedure at his earliest convenience. The implantable loop recorder will be interrogated at least once a month for up to 12 months to retrieve the information that has been recorded during their hemodialysis treatment. During this time, the patient participant will complete a questionnaire too using the LEVIL application. Then, 12 months after the initial insertion of the device, a follow-up call will be completed by a member of the research team where the patient will have the choice to have the device removed if desired. If the patient chooses to keep the device, we will monitor the implantable loop recorder for another year and the patient will be transferred to LHSC's Inherited Heart Rhythm Clinic at University Hospital for clinical monitoring after this. Completion of the questionnaire will continue during this time. If they choose to have the device removed, the cardiac electrophysiologist will remove the device at his earliest convenience.

Bloodwork will be obtained pre and post dialysis as well as at peak stress of each imaging session. This will allow us to assess for relevant biomarkers of oxidative stress, myocardial ischemia, and volume overload.

ELIGIBILITY:
Inclusion Criteria:

* No significant residual renal function (<250ml of urine per day).
* Must be on hemodialysis for at least 3 months
* Age ≥18 years
* Able/willing to provide informed consent

Exclusion Criteria:

* Presence of a pacemaker and implantable cardioverter defibrillator
* Prior diagnosis of chronic arrhythmia and/or are on anti-arrhythmic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Temporal association between dialysis induced cardiac injury and frequency of arrhythmia | Through heart monitoring of 12 months
  The primary outcome will be to determine the correlation between dialysis cardiac injury and the rate of arrhythmia. This will be measured by comparing perfusion heterogeneity in CT images to the rhythms recorded on the Reveal LINQ heart monitor.
Temporal association between dialysis induced cardiac injury and electrophysiological substrate responsible for arrhythmia. | Through imaging session, on average of 4 hours
  The primary outcome will be to determine the correlation between dialysis cardiac injury and the electrophysiological substrate responsible for arrhythmia. This will be measured by comparing perfusion heterogeneity in CT images to the results of the electrophysiological maps.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W McIntyre, MD, Principal Investigator — London Health Sciences Centre
Locations (2):
- Canada (2):
  - University Hospital, London, Ontario
  - Kidney Care Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No